CLINICAL TRIAL: NCT02654002
Title: A Phase 1 Study in Healthy Volunteers to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of GS-9674, and the Effect of Food on GS-9674 Pharmacokinetics and Pharmacodynamics
Brief Title: Study in Healthy Volunteers to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of GS-9674 (Cilofexor), and the Effect of Food on GS-9674 Pharmacokinetics and Pharmacodynamics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-402-1851
Record Dates: First submitted 2016-01-11; First posted 2016-01-13 (Estimated); Results first posted 2020-10-12 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-09

CONDITIONS: Nonalcoholic Steatohepatitis (NASH)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — cilofexor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Cohort 1: Cilofexor 10 mg (Experimental): Participants in fasted state will receive cilofexor 10 mg or placebo once on Day 1 followed by a 5-day washout period then receive cilofexor 10 mg or placebo once daily from Day 7 to Day 20.
  Interventions: Drug: Cilofexor; Drug: Placebo
- Cohort 2: Cilofexor 30 mg (Experimental): Participants in fasted state will receive cilofexor 30 mg or placebo once on Day 1 followed by a 5-day washout period then receive cilofexor 30 mg or placebo once daily from Day 7 to Day 20.
  Interventions: Drug: Cilofexor; Drug: Placebo
- Cohort 3: Cilofexor 100 mg (Experimental): Participants in fasted state will receive cilofexor 100 mg or placebo once on Day 1 followed by a 5-day washout period then receive cilofexor 100 mg or placebo once daily from Day 7 to Day 20.
  Interventions: Drug: Cilofexor; Drug: Placebo
- Cohort 4: Cilofexor 300 mg (Experimental): Participants in fasted state will receive cilofexor 300 mg or placebo once on Day 1 followed by a 5-day washout period then receive cilofexor 300 mg or placebo once daily from Day 7 to Day 20.
  Interventions: Drug: Cilofexor; Drug: Placebo
- Cohort 5: Cilofexor 100 mg (Experimental): Participants in fed state will receive cilofexor 100 mg or placebo once with food on Day 1 followed by a 5-day washout period then receive cilofexor 100 mg or placebo tablet, orally, once daily with food from Day 7 to Day 20.
  Interventions: Drug: Cilofexor; Drug: Placebo
- Cohort 6: Cilofexor 50 mg (Experimental): Participants in fed state will receive cilofexor 50 mg or placebo twice with food on Day 1 followed by a 5-day washout period then receive cilofexor 50 mg or placebo twice daily from Day 7 to Day 20.
  Interventions: Drug: Cilofexor; Drug: Placebo
- Cohort 7: Cilofexor 15 mg (Experimental): Participants in fed state will receive cilofexor 15 mg or placebo twice with food on Day 1 followed by a 5-day washout period then receive cilofexor 15 mg or placebo twice daily from Day 7 to Day 20.
  Interventions: Drug: Cilofexor; Drug: Placebo
- Cohort 8: Cilofexor 10 mg (Experimental): Participants in fed state will receive cilofexor 10 mg or placebo once with food on Day 1 followed by a 5-day washout period then receive cilofexor 10 mg or placebo once daily from Day 7 to Day 20.
  Interventions: Drug: Cilofexor; Drug: Placebo
- Cohort 9: Cilofexor (Experimental): Participants will receive cilofexor up to 300 mg or placebo once daily in the evening on empty stomach.
  Interventions: Drug: Cilofexor; Drug: Placebo
- Cohort 10: Cilofexor (Experimental): Participants will receive cilofexor up to 300 mg or placebo once daily in the evening on empty stomach.
  Interventions: Drug: Cilofexor; Drug: Placebo

INTERVENTIONS:
Drug: Cilofexor — Tablets administered orally
  Other Names: GS-9674
Drug: Placebo — Tablets administered orally

SUMMARY:
This study will evaluate the safety and tolerability of escalating single- and multiple-oral doses of cilofexor, and characterize the single- and multiple-dose pharmacokinetics (PK) of cilofexor. The study will be conducted in 3 parts (Part A, Part B, and Part C). Participants will receive either cilofexor or cilofexor placebo.

Part A will proceed in 4 prespecified staggered cohorts. Within each cohort, the cumulative, blinded safety data will be evaluated for dose escalation from single-dose (Period 1) to multiple-dose (Period 2). Based on the available safety, pharmacokinetics, and/or pharmacodynamics (PD) data from cohorts in Part A and Part C (if applicable), total daily doses and frequency of dosing will be chosen for the cohorts in Part B. Parts B and C will consist of adaptive cohorts and may be initiated in parallel. Part B cohorts may be initiated in parallel with cohorts in Part A if the total dose under evaluation is at or below a dose already evaluated.

This study is partially blinded (no one is blinded on Day -1).

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy male and non-pregnant, non-lactating female volunteers
* Body mass index (BMI) 19 ≤ BMI ≤ 30 kg/m^2
* Normal 12-lead electrocardiogram (ECG) or one with abnormalities that are considered clinically insignificant by the investigator
* Normal renal function (estimated glomerular filtration rate calculated using the Cockcroft-Gault equation ≥ 80 mL/min)
* No significant medical history, and in good general health as determined by the investigator at screening evaluation performed no more than 28 days prior to the scheduled first dose.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2016-01-20 (Actual); Primary Completion 2016-07-14 (Actual); Study Completion 2016-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (1):
- SeaView Research, Inc, Miami, Florida, United States

REFERENCES:
- [Background] Djedjos CS, Kirby BJ, Billin A, Gosink J, Song Q, Srihari R, et al. Pharmacodynamic Effects of the Oral, Non-Steroidal Farnesoid X Receptor Agonist GS-9674 in Healthy Volunteers. The 67th Annual Meeting of the American Association for the Study of Liver Diseases: The Liver Meeting (AASLD); 2016 November 11-15; Boston MA United States.
- [Background] Kirby BJ, Djedjos CS, Birkeback J, Song Q, Grycz K, Weston J, et al. Evaluation of the Safety and Pharmacokinetics of the Oral, Nonsteroidal Farnesoid X Receptor Agonist GS-9674 in Healthy Volunteers. The 67th Annual Meeting of the American Association for the Study of Liver Diseases: The Liver Meeting (AASLD); 2016 November 11-15; Boston MA United States.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at one study site in the United States. The first participant was screened on 20 January 2016. The last study visit occurred on 14 July 2016.
Pre-assignment Details: 183 participants were screened. No participants were enrolled in Cohorts 9 and 10.
Groups:
- Cohort 1: Cilofexor 10 mg: Participants in fasted state received cilofexor 10 mg tablet, orally, once on Day 1 followed by a 5-day washout period then received cilofexor 10 mg tablet, orally, once daily from Day 7 to Day 20.
- Cohort 2: Cilofexor 30 mg: Participants in fasted state received cilofexor 30 mg tablet, orally, once on Day 1 followed by a 5-day washout period then received cilofexor 30 mg tablet, orally, once daily from Day 7 to Day 20.
- Cohort 3: Cilofexor 100 mg: Participants in fasted state received cilofexor 100 mg tablet, orally, once on Day 1 followed by a 5-day washout period then received cilofexor 100 mg tablet, orally, once daily from Day 7 to Day 20.
- Cohort 4: Cilofexor 300 mg: Participants in fasted state received cilofexor 300 mg tablet, orally, once on Day 1 followed by a 5-day washout period then received cilofexor 300 mg tablet, orally, once daily from Day 7 to Day 20.
- Cohort 5: Cilofexor 100 mg: Participants in fed state received cilofexor 100 mg tablet, orally, once with food on Day 1 followed by a 5-day washout period then received cilofexor 100 mg tablet, orally, once daily with food from Day 7 to Day 20.
- Cohort 6: Cilofexor 50 mg: Participants in fed state received cilofexor 50 mg tablet, orally, twice with food on Day 1 followed by a 5-day washout period then received cilofexor 50 mg tablet, orally, twice daily from Day 7 to Day 20.
- Cohort 7: Cilofexor 15 mg: Participants in fed state received cilofexor 15 mg tablet orally, twice with food on Day 1 followed by a 5-day washout period then received cilofexor 15 mg tablet orally, twice daily from Day 7 to Day 20.
- Cohort 8: Cilofexor 10 mg: Participants in fed state received cilofexor 10 mg tablet, orally, once with food on Day 1 followed by a 5-day washout period then received cilofexor 10 mg tablet, orally, once daily from Day 7 to Day 20.
- All Placebo: Participants in fasted state (cohorts 1-4) and fed state (cohorts 5-8) received placebo tablet(s), orally, once or twice on Day 1 followed by a 5-day washout period then received placebo tablet(s), orally, once or twice daily from Day 7 to Day 20.
Period: Overall Study
Arm/Group | Cohort 1: Cilofexor 10 mg | Cohort 2: Cilofexor 30 mg | Cohort 3: Cilofexor 100 mg | Cohort 4: Cilofexor 300 mg | Cohort 5: Cilofexor 100 mg | Cohort 6: Cilofexor 50 mg | Cohort 7: Cilofexor 15 mg | Cohort 8: Cilofexor 10 mg | All Placebo
Started | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 24
Completed | 12 | 12 | 12 | 12 | 12 | 11 | 11 | 11 | 24
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrew Consent | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all randomized participants who took at least 1 dose of study drug. Participants were grouped according to the treatment they actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Cilofexor 10 mg | Cohort 2: Cilofexor 30 mg | Cohort 3: Cilofexor 100 mg | Cohort 4: Cilofexor 300 mg | Cohort 5: Cilofexor 100 mg | Cohort 6: Cilofexor 50 mg | Cohort 7: Cilofexor 15 mg | Cohort 8: Cilofexor 10 mg | All Placebo | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 11 | 12 | 11 | 24 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (6.5) | 35 (8.9) | 37 (6.1) | 32 (8.7) | 40 (4.6) | 33 (7.4) | 35 (6.0) | 35 (7.1) | 36 (6.7) | 35 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 5 | 4 | 5 | 6 | 7 | 8 | 14 | 59
  Male | 6 | 8 | 7 | 8 | 7 | 5 | 5 | 3 | 10 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 12 | 11 | 12 | 12 | 11 | 12 | 11 | 24 | 116
  Not Hispanic or Latino | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black | 1 | 1 | 2 | 3 | 2 | 2 | 1 | 2 | 2 | 16
  Race: White | 11 | 11 | 10 | 9 | 10 | 9 | 11 | 9 | 22 | 102
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 12 | 12 | 12 | 11 | 12 | 11 | 24 | 118

OUTCOME MEASURES:

1. Primary Outcome: Single-Dose Pharmacokinetic (PK) Parameter: AUClast of Cilofexor
Description: AUClast is defined as the concentration of drug from time zero to the last quantifiable concentration.
Time Frame: Day 1: -0.5, 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 16, 24, 48, 72, and 96 hours post-dose
Population: The PK Analysis Set included all randomized participants who took at least 1 dose of Cilofexor and had at least 1 non-missing post-dose concentration value reported by the PK laboratory for each corresponding analyte.
Measure: Mean (Standard Deviation); unit: hours*nanogram/millilitre (h*ng/mL)
Arm/Group | Cohort 1: Cilofexor 10 mg | Cohort 2: Cilofexor 30 mg | Cohort 3: Cilofexor 100 mg | Cohort 4: Cilofexor 300 mg | Cohort 5: Cilofexor 100 mg | Cohort 6: Cilofexor 50 mg | Cohort 7: Cilofexor 15 mg | Cohort 8: Cilofexor 10 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 11 | 12 | 11
hours*nanogram/millilitre (h*ng/mL) | 1236.0 (384.65) | 2450.6 (921.70) | 7712.1 (7270.76) | 12458.8 (4223.12) | 4979.5 (2039.07) | 3091.4 (752.66) | 1301.9 (388.51) | 905.9 (210.24)

2. Primary Outcome: Single-Dose PK Parameter: AUCinf of Cilofexor
Description: AUCinf is defined as the concentration of drug extrapolated to infinite time (area under the plasma concentration versus time curve extrapolated to infinite time).
Time Frame: as for outcome 1
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Cohort 1: Cilofexor 10 mg | Cohort 2: Cilofexor 30 mg | Cohort 3: Cilofexor 100 mg | Cohort 4: Cilofexor 300 mg | Cohort 5: Cilofexor 100 mg | Cohort 6: Cilofexor 50 mg | Cohort 7: Cilofexor 15 mg | Cohort 8: Cilofexor 10 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 11 | 12 | 11
h*ng/mL | 1255.9 (382.37) | 2473.4 (920.85) | 7743.7 (7273.50) | 12495.7 (4230.00) | 5016.7 (2022.94) | 3559.2 (1092.73) | 1409.3 (428.33) | 924.0 (216.60)

3. Primary Outcome: Single-Dose PK Parameter: Cmax of Cilofexor
Description: Cmax is defined as the maximum observed concentration of drug in plasma.
Time Frame: as for outcome 1
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: Cilofexor 10 mg | Cohort 2: Cilofexor 30 mg | Cohort 3: Cilofexor 100 mg | Cohort 4: Cilofexor 300 mg | Cohort 5: Cilofexor 100 mg | Cohort 6: Cilofexor 50 mg | Cohort 7: Cilofexor 15 mg | Cohort 8: Cilofexor 10 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 11 | 12 | 11
ng/mL | 304.2 (126.66) | 580.2 (283.79) | 2592.3 (3059.31) | 3055.5 (2022.27) | 927.6 (540.94) | 665.9 (152.30) | 340.2 (124.44) | 209.8 (63.24)

4. Primary Outcome: Multiple-Dose PK Parameter: AUCtau of Cilofexor
Description: AUCtau is the concentration of drug over time (area under the plasma concentration versus time curve over the dosing interval).
Time Frame: Day 20: -0.5, 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 16, 24, 48, 72, and 96 hours post-dose
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Cohort 1: Cilofexor 10 mg | Cohort 2: Cilofexor 30 mg | Cohort 3: Cilofexor 100 mg | Cohort 4: Cilofexor 300 mg | Cohort 5: Cilofexor 100 mg | Cohort 6: Cilofexor 50 mg | Cohort 7: Cilofexor 15 mg | Cohort 8: Cilofexor 10 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 11 | 11 | 11
h*ng/mL | 1284.9 (460.35) | 2891.0 (680.10) | 6719.4 (3980.90) | 8486.0 (4139.86) | 4182.7 (1956.03) | 3698.3 (837.91) | 1293.5 (250.95) | 848.2 (213.82)

5. Primary Outcome: Multiple-Dose PK Parameter: Cmax of Cilofexor
Description: Cmax is defined as the maximum observed concentration of drug in plasma.
Time Frame: as for outcome 4
Population: Participants in the PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: Cilofexor 10 mg | Cohort 2: Cilofexor 30 mg | Cohort 3: Cilofexor 100 mg | Cohort 4: Cilofexor 300 mg | Cohort 5: Cilofexor 100 mg | Cohort 6: Cilofexor 50 mg | Cohort 7: Cilofexor 15 mg | Cohort 8: Cilofexor 10 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 11 | 11 | 11
ng/mL | 322.2 (136.70) | 717.5 (235.50) | 2231.2 (1693.78) | 2327.9 (1897.48) | 818.7 (437.28) | 697.8 (145.60) | 290.4 (78.71) | 187.0 (57.10)

6. Primary Outcome: Multiple-Dose PK Parameter: Ctau of Cilofexor
Description: Ctau is defined as the observed drug concentration at the end of the dosing interval.
Time Frame: as for outcome 4
Population: Participants in the PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: Cilofexor 10 mg | Cohort 2: Cilofexor 30 mg | Cohort 3: Cilofexor 100 mg | Cohort 4: Cilofexor 300 mg | Cohort 5: Cilofexor 100 mg | Cohort 6: Cilofexor 50 mg | Cohort 7: Cilofexor 15 mg | Cohort 8: Cilofexor 10 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 11 | 11 | 11
ng/mL | 2.7 (1.53) | 7.9 (3.97) | 36.3 (15.44) | 70.1 (39.46) | 22.6 (8.44) | 107.6 (84.58) | 28.4 (14.13) | 3.0 (1.54)

7. Primary Outcome: Percentage of Participants With at Least One Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant administered a medicinal product, which does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and/or unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: First dose date up to last dose date (Maximum: 20 days) plus 30 days
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Cilofexor 10 mg | Cohort 2: Cilofexor 30 mg | Cohort 3: Cilofexor 100 mg | Cohort 4: Cilofexor 300 mg | Cohort 5: Cilofexor 100 mg | Cohort 6: Cilofexor 50 mg | Cohort 7: Cilofexor 15 mg | Cohort 8: Cilofexor 10 mg | All Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 11 | 12 | 11 | 24
percentage of participants | 33.3 | 25.0 | 33.3 | 25.0 | 41.7 | 27.3 | 75.0 | 18.2 | 29.2

8. Primary Outcome: Percentage of Participants With Clinically Significant 12-Lead Electrocardiogram (ECG) Abnormalities
Description: Investigator determined the ECG findings were clinically significant.
Time Frame: First dose date up to last dose date (Maximum: 20 days) plus 30 days
Population: Participants in the Safety Analysis Set were analyzed. Participants were grouped according to the treatment they actually received.
Measure: Number; unit: percentage of participants
Groups:
- Cohort 1: Cilofexor 10 mg: Participants in fasted state received cilofexor 10 mg tablet, orally, once on Day 1 followed by a 5-day washout period then receive cilofexor 10 mg tablet, orally, once daily from Day 7 to Day 20.
- Cohort 2: Cilofexor 30 mg: Participants in fasted state received cilofexor 30 mg tablet, orally, once on Day 1 followed by a 5-day washout period then receive cilofexor 30 mg tablet, orally, once daily from Day 7 to Day 20.
- Cohort 3: Cilofexor 100 mg: Participants in fasted state received cilofexor 100 mg tablet, orally, once on Day 1 followed by a 5-day washout period then receive cilofexor 100 mg tablet, orally, once daily from Day 7 to Day 20.
- Cohort 4: Cilofexor 300 mg: Participants in fasted state received cilofexor 300 mg tablet, orally, once on Day 1 followed by a 5-day washout period then receive cilofexor 300 mg tablet, orally, once daily from Day 7 to Day 20.
- Cohort 5: Cilofexor 100 mg: Participants in fed state received cilofexor 100 mg tablet, orally, once with food on Day 1 followed by a 5-day washout period then receive cilofexor 100 mg tablet, orally, once daily with food from Day 7 to Day 20.
- Cohort 6: Cilofexor 50 mg: Participants in fed state received cilofexor 50 mg tablet, orally, twice with food on Day 1 followed by a 5-day washout period then receive cilofexor 50 mg tablet, orally, twice daily from Day 7 to Day 20.
- Cohort 7: Cilofexor 15 mg: Participants in fed state received cilofexor 15 mg tablet orally, twice with food on Day 1 followed by a 5-day washout period then receive cilofexor 15 mg tablet orally, twice daily from Day 7 to Day 20.
- Cohort 8: Cilofexor 10 mg: Participants in fed state received cilofexor 10 mg tablet, orally, once with food on Day 1 followed by a 5-day washout period then receive cilofexor 10 mg tablet, orally, once daily from Day 7 to Day 20.
- All Placebo: Participants in fasted state (cohorts 1-4) and fed state (cohorts 5-8) received placebo tablet(s), orally, once or twice on Day 1 followed by a 5-day washout period then receive placebo tablet(s), orally, once or twice daily from Day 7 to Day 20.
Arm/Group | Cohort 1: Cilofexor 10 mg | Cohort 2: Cilofexor 30 mg | Cohort 3: Cilofexor 100 mg | Cohort 4: Cilofexor 300 mg | Cohort 5: Cilofexor 100 mg | Cohort 6: Cilofexor 50 mg | Cohort 7: Cilofexor 15 mg | Cohort 8: Cilofexor 10 mg | All Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 11 | 12 | 11 | 24
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Percentage of Participants With Clinical Laboratory Abnormalities
Description: Treatment-emergent laboratory (Hematology, Chemistry, and Urinalysis) abnormalities were defined as values that increase at least one toxicity grade from baseline. Laboratory Abnormalities are graded by the investigator as Grade 1, 2, 3, or 4 according to the modified Gilead Sciences, Inc (GSI) Grading Scale. The most severe graded abnormality from all tests was counted for each participant. Data is only reported for those Grades reported in 1 or more participants.
Time Frame: First dose date up to last dose date (Maximum: 20 days) plus 30 days
Population: Participants in the Safety Analysis Set with available data were analyzed. Participants were grouped according to the treatment they actually received.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Cilofexor 10 mg | Cohort 2: Cilofexor 30 mg | Cohort 3: Cilofexor 100 mg | Cohort 4: Cilofexor 300 mg | Cohort 5: Cilofexor 100 mg | Cohort 6: Cilofexor 50 mg | Cohort 7: Cilofexor 15 mg | Cohort 8: Cilofexor 10 mg | All Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 11 | 12 | 11 | 24
percentage of participants
  Activated Partial Thromboplastin Time: Grade 1 | 0.0 | 8.3 | 16.7 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Hemoglobin-Hypo: Grade 1 | 16.7 | 25.0 | 16.7 | 8.3 | 16.7 | 18.2 | 25.0 | 27.3 | 29.2
  Hemoglobin-Hypo: Grade 2 | 0.0 | 0.0 | 8.3 | 8.3 | 8.3 | 0.0 | 16.7 | 9.1 | 8.3
  Hemoglobin-Hypo: Grade 3 | 0.0 | 0.0 | 0.0 | 8.3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  International Normalized Ratio: Grade 2 | 0.0 | 0.0 | 0.0 | 0.0 | 8.3 | 0.0 | 0.0 | 0.0 | 0.0
  Lymphocytes: Grade 1 | 0.0 | 8.3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Platelets: Grade 2 | 0.0 | 8.3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Alanine Aminotransferase: Grade 1 | 0.0 | 0.0 | 0.0 | 8.3 | 0.0 | 0.0 | 0.0 | 9.1 | 4.2
  Alanine Aminotransferase: Grade 2 | 0.0 | 16.7 | 0.0 | 0.0 | 8.3 | 9.1 | 0.0 | 0.0 | 4.2
  Alanine Aminotransferase: Grade 3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 8.3 | 0.0 | 0.0
  Aspartate Aminotransferase: Grade 1 | 0.0 | 0.0 | 0.0 | 0.0 | 8.3 | 9.1 | 0.0 | 0.0 | 4.2
  Aspartate Aminotransferase: Grade 2 | 0.0 | 8.3 | 0.0 | 0.0 | 0.0 | 0.0 | 8.3 | 0.0 | 0.0
  Aspartate Aminotransferase: Grade 3 | 0.0 | 8.3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Aspartate Aminotransferase: Grade 4 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 4.2
  Albumin Corrected Calcium-Hyper: Grade 1 | 0.0 | 0.0 | 0.0 | 8.3 | 8.3 | 9.1 | 8.3 | 0.0 | 4.2
  Gamma-Glutamyltransferase: Grade 1 | 0.0 | 0.0 | 8.3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 4.2
  Gamma-Glutamyltransferase: Grade 2 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 8.3 | 0.0 | 0.0
  Low-Density Lipoprotein: Grade 1 | 8.3 | 0.0 | 8.3 | 8.3 | 25.0 | 27.3 | 25.0 | 18.2 | 12.5
  Low-Density Lipoprotein: Grade 2 | 8.3 | 8.3 | 8.3 | 8.3 | 16.7 | 0.0 | 8.3 | 0.0 | 4.2
  Phosphate-Hypo: Grade 1 | 0.0 | 8.3 | 0.0 | 8.3 | 8.3 | 0.0 | 8.3 | 9.1 | 4.2
  Phosphate-Hypo: Grade 2 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 4.2
  Serum Amylase: Grade 1 | 0.0 | 8.3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Serum Amylase: Grade 2 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 9.1 | 4.2
  Serum Glucose,Fasting-Hyper: Grade 1 | 0.0 | 8.3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Serum Glucose,Fasting-Hyper:Grade 2 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 9.1 | 0.0
  Serum Glucose,Non-Fasting-Hyper:Grade 1: number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 11 | 11 | 11 | 24
  Serum Glucose,Non-Fasting-Hyper:Grade 1 | 0.0 | 0.0 | 0.0 | 0.0 | 58.3 | 0.0 | 18.2 | 0.0 | 4.2
  Serum Glucose,Non-Fasting-Hyper:Grade 2: number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 11 | 11 | 11 | 24
  Serum Glucose,Non-Fasting-Hyper:Grade 2 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 9.1 | 0.0
  Serum Glucose,Non-Fasting-Hypo:Grade 1 | 0.0 | 0.0 | 0.0 | 0.0 | 8.3 | 0.0 | 0.0 | 0.0 | 4.2
  Serum Potassium-Hypo:Grade 1 | 0.0 | 8.3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 27.3 | 0.0
  Serum Sodium-Hyper:Grade 1 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 9.1 | 0.0
  Serum Sodium-Hypo:Grade 1 | 8.3 | 25.0 | 8.3 | 0.0 | 0.0 | 18.2 | 50.0 | 9.1 | 4.2
  Total Bilirubin-Hyper:Grade 1 | 0.0 | 0.0 | 0.0 | 8.3 | 0.0 | 0.0 | 0.0 | 9.1 | 4.2
  Total Cholesterol-Hyper:Grade 1 | 16.7 | 0.0 | 16.7 | 16.7 | 25.0 | 36.4 | 25.0 | 9.1 | 12.5
  Total Cholesterol-Hyper:Grade 2 | 8.3 | 0.0 | 8.3 | 0.0 | 16.7 | 0.0 | 8.3 | 9.1 | 4.2
  Uric Acid-Hyper:Grade 1 | 0.0 | 0.0 | 8.3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Uric Acid-Hypo:Grade 1 | 8.3 | 16.7 | 0.0 | 8.3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Occult Blood: Grade 1 | 0.0 | 0.0 | 8.3 | 0.0 | 8.3 | 0.0 | 0.0 | 9.1 | 8.3
  Occult Blood: Grade 2 | 16.7 | 8.3 | 0.0 | 8.3 | 0.0 | 0.0 | 0.0 | 9.1 | 12.5
  Occult Blood: Grade 3 | 25.0 | 8.3 | 8.3 | 16.7 | 8.3 | 18.2 | 16.7 | 18.2 | 8.3
  Urine Glucose: Grade 1 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 9.1 | 0.0
  Urine Protein: Grade 1 | 0.0 | 8.3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 4.2

10. Secondary Outcome: Pharmacodynamic (PD) Parameter: Fibroblast Growth Factor 19 (FGF19) AUC2-12 Ratio
Description: AUC2-12 is defined as the AUC from time 2 to 12 hours. The ratios calculated were normalized to Day -1. Participants received a single placebo tablet at Day -1 for Baseline. The ratio reported for Day 1 is the AUC2-12 Day 1 /AUC2-12 Day-1. The ratio reported for Day 20 is the AUC2-12 Day 20 /AUC2-12 Day-1.
Time Frame: Day -1: -0.5, 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, and 16 hours post-dose; Days 1, and 20: -0.5, 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 16, 24, 48, 72, and 96 hours post-dose
Population: The PD Analysis Set included all randomized participants who received at least 1 dose of study drug and had the necessary baseline and on-study measurement to provide interpretable results for each respective PD parameter. Included participants with available data.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Groups:
- All Fasted Placebo: Participants in fasted state (cohorts 1-4) received placebo tablet(s), orally, once on Day 1 followed by a 5-day washout period then received placebo tablet(s), orally, once daily from Day 7 to Day 20.
- All Fed Placebo: Participants in fed state (cohorts 5-8) received placebo tablet(s), orally, once or twice on Day 1 followed by a 5-day washout period then received placebo tablet(s), orally, once or twice daily from Day 7 to Day 20.
Arm/Group | Cohort 1: Cilofexor 10 mg | Cohort 2: Cilofexor 30 mg | Cohort 3: Cilofexor 100 mg | Cohort 4: Cilofexor 300 mg | All Fasted Placebo | Cohort 5: Cilofexor 100 mg | Cohort 6: Cilofexor 50 mg | Cohort 7: Cilofexor 15 mg | Cohort 8: Cilofexor 10 mg | All Fed Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 11 | 12 | 11 | 12
ratio
  Day 1/Day -1 | 2.040 [1.571 to 2.650] | 1.958 [1.478 to 2.594] | 2.037 [1.699 to 2.442] | 2.314 [1.958 to 2.735] | 0.981 [0.777 to 1.240] | 2.406 [2.196 to 2.637] | 2.629 [2.369 to 2.917] | 1.743 [1.463 to 2.076] | 1.372 [1.132 to 1.663] | 0.916 [0.799 to 1.050]
  Day 20/Day -1: number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 11 | 11 | 11 | 12
  Day 20/Day -1 | 2.270 [1.500 to 3.435] | 2.261 [1.782 to 2.868] | 2.054 [1.727 to 2.442] | 2.179 [1.632 to 2.911] | 1.249 [0.929 to 1.681] | 1.795 [1.544 to 2.086] | 2.119 [1.728 to 2.598] | 1.650 [1.301 to 2.093] | 1.509 [1.325 to 1.719] | 0.963 [0.762 to 1.216]

11. Secondary Outcome: PD Parameter: FGF19 Cmax Ratio
Description: Cmax is defined as the maximum observed concentration of FGF19 in plasma. The ratios calculated were normalized to Day -1. Participants received a single placebo tablet at Day -1 for Baseline. The ratio reported for Day 1 is the Cmax Day 1 /Cmax Day-1. The ratio reported for Day 20 is the Cmax Day 20 /Cmax Day-1.
Time Frame: as for outcome 10
Population: Participants in the PD Analysis Set with available data were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Cohort 1: Cilofexor 10 mg | Cohort 2: Cilofexor 30 mg | Cohort 3: Cilofexor 100 mg | Cohort 4: Cilofexor 300 mg | All Fasted Placebo | Cohort 5: Cilofexor 100 mg | Cohort 6: Cilofexor 50 mg | Cohort 7: Cilofexor 15 mg | Cohort 8: Cilofexor 10 mg | All Fed Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 11 | 12 | 11 | 12
ratio
  Day 1/Day -1 | 2.217 [1.667 to 2.949] | 2.084 [1.468 to 2.957] | 2.259 [1.742 to 2.930] | 2.679 [2.113 to 3.398] | 0.982 [0.759 to 1.272] | 2.793 [2.264 to 3.446] | 2.973 [2.578 to 3.428] | 1.961 [1.588 to 2.422] | 1.689 [1.354 to 2.106] | 0.929 [0.810 to 1.065]
  Day 20/Day -1: number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 11 | 11 | 11 | 12
  Day 20/Day -1 | 2.157 [1.345 to 3.460] | 2.393 [1.770 to 3.235] | 2.325 [1.804 to 2.996] | 3.084 [2.194 to 4.334] | 1.210 [0.910 to 1.608] | 2.241 [1.850 to 2.713] | 2.455 [1.964 to 3.069] | 1.768 [1.270 to 2.462] | 1.878 [1.527 to 2.310] | 0.874 [0.680 to 1.123]

12. Secondary Outcome: PD Parameter: 7alpha-hydroxy-4-cholesten-3-one (C4) AUC2-12 Ratio
Description: as for outcome 10
Time Frame: as for outcome 10
Population: Participants in the PD Analysis Set with available data were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Cohort 1: Cilofexor 10 mg | Cohort 2: Cilofexor 30 mg | Cohort 3: Cilofexor 100 mg | Cohort 4: Cilofexor 300 mg | All Fasted Placebo | Cohort 5: Cilofexor 100 mg | Cohort 6: Cilofexor 50 mg | Cohort 7: Cilofexor 15 mg | Cohort 8: Cilofexor 10 mg | All Fed Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 11 | 12 | 11 | 12
ratio
  Day 1/Day -1 | 0.681 [0.431 to 1.077] | 0.640 [0.516 to 0.794] | 0.427 [0.340 to 0.537] | 0.347 [0.278 to 0.433] | 1.147 [0.921 to 1.429] | 0.837 [0.629 to 1.114] | 0.653 [0.581 to 0.735] | 0.863 [0.747 to 0.997] | 1.108 [0.828 to 1.483] | 1.057 [0.893 to 1.252]
  Day 20/Day -1: number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 11 | 11 | 11 | 12
  Day 20/Day -1 | 0.661 [0.456 to 0.959] | 0.382 [0.277 to 0.525] | 0.495 [0.348 to 0.704] | 0.325 [0.223 to 0.474] | 1.213 [0.828 to 1.777] | 0.621 [0.414 to 0.933] | 0.173 [0.109 to 0.275] | 0.624 [0.472 to 0.825] | 0.974 [0.677 to 1.402] | 0.843 [0.681 to 1.043]

13. Secondary Outcome: PD Parameter: C4 Cmin Ratio
Description: Cmin is defined as the minimum observed concentration of C4 in plasma. The ratios calculated were normalized to Day -1. Participants received a single placebo tablet at Day -1 for Baseline. The ratio reported for Day 1 is the Cmin Day 1 /Cmin Day-1. The ratio reported for Day 20 is the Cmin Day 20 /Cmin Day-1.
Time Frame: as for outcome 10
Population: Participants in the PD Analysis Set with available data were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Cohort 1: Cilofexor 10 mg | Cohort 2: Cilofexor 30 mg | Cohort 3: Cilofexor 100 mg | Cohort 4: Cilofexor 300 mg | All Fasted Placebo | Cohort 5: Cilofexor 100 mg | Cohort 6: Cilofexor 50 mg | Cohort 7: Cilofexor 15 mg | Cohort 8: Cilofexor 10 mg | All Fed Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 11 | 12 | 11 | 12
ratio
  Day 1/Day -1 | 0.715 [0.531 to 0.964] | 0.759 [0.597 to 0.964] | 0.663 [0.542 to 0.810] | 0.467 [0.370 to 0.589] | 1.201 [0.941 to 1.532] | 0.613 [0.497 to 0.756] | 0.348 [0.260 to 0.467] | 0.737 [0.590 to 0.921] | 0.961 [0.787 to 1.173] | 1.162 [0.981 to 1.377]
  Day 20/Day -1: number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 11 | 11 | 11 | 12
  Day 20/Day -1 | 0.822 [0.580 to 1.163] | 0.456 [0.303 to 0.687] | 0.624 [0.458 to 0.850] | 0.432 [0.277 to 0.675] | 1.262 [0.901 to 1.767] | 0.440 [0.264 to 0.733] | 0.116 [0.071 to 0.192] | 0.508 [0.334 to 0.773] | 0.862 [0.666 to 1.115] | 0.983 [0.718 to 1.346]

ADVERSE EVENTS:
Time Frame: First dose date up to last dose date (Maximum: 20 days) plus 30 days
Description: The Safety Analysis Set included all randomized participants who took at least 1 dose of study drug. Participants were grouped according to the treatment they actually received.
Arm/Group | Cohort 1: Cilofexor 10 mg | Cohort 2: Cilofexor 30 mg | Cohort 3: Cilofexor 100 mg | Cohort 4: Cilofexor 300 mg | Cohort 5: Cilofexor 100 mg | Cohort 6: Cilofexor 50 mg | Cohort 7: Cilofexor 15 mg | Cohort 8: Cilofexor 10 mg | All Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/11 | 0/12 | 0/11 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/11 | 0/12 | 0/11 | 0/24
Other Adverse Events (participants affected / at risk) | 4/12 | 3/12 | 4/12 | 3/12 | 5/12 | 3/11 | 9/12 | 2/11 | 6/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Cilofexor 10 mg (N=12) | Cohort 2: Cilofexor 30 mg (N=12) | Cohort 3: Cilofexor 100 mg (N=12) | Cohort 4: Cilofexor 300 mg (N=12) | Cohort 5: Cilofexor 100 mg (N=12) | Cohort 6: Cilofexor 50 mg (N=11) | Cohort 7: Cilofexor 15 mg (N=12) | Cohort 8: Cilofexor 10 mg (N=11) | All Placebo (N=24)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1
Ocular discomfort (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 5 | 0 | 3
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years